CLINICAL TRIAL: NCT06972433
Title: Comparison of Endodontic Flare up in Single Visit Root Canal Treatment Versus Multiple Visit Root Canal Treatment in Patients Visiting Scd, Swat.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Warisha Ubaid, trainee medical officer at saidu college of dentistry ,swat, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106-ERB/024
Record Dates: First submitted 2025-05-13; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Complication; Root Canal Therapy; Pulpitis - Irreversible
Keywords: enddoontic flare-ups, root canal therapy, single visit root canal treatment, multiple visit root canal treatment
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only the participant will be blinded to the group assignment (single-visit vs. multiple-visit root canal treatment). The care provider and investigator will be aware of the allocation due to procedural differences. Blinding of participants is maintained by not informing them about the number of treatment visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single visit root canal treatment (Experimental): Patients receive complete root canal therapy in a single appointment, including cleaning, shaping, and obturation of canals.
  Interventions: Procedure: single visit root canal treatment
- Multiple visit root canal treatment (Active Comparator): Patients receive root canal therapy over multiple appointments, with canal medication between visits before final obturation.
  Interventions: Procedure: Multiple visit root canal treatment

INTERVENTIONS:
Procedure: single visit root canal treatment — Root canal procedure performed in a single visit using ProTaper file system, sodium hypochlorite irrigation, and lateral compaction with gutta-percha and sealer. Final restoration with GIC.
  Arms: Single visit root canal treatment
Procedure: Multiple visit root canal treatment — Root canal procedure performed over two or more visits using the same instrumentation and irrigation protocol. Canals are medicated between appointments before obturation and restoration.
  Arms: Multiple visit root canal treatment

SUMMARY:
This randomized controlled trial aims to compare the incidence of endodontic flare-ups in patients undergoing single-visit versus multiple-visit root canal treatment (RCT) at Saidu College of Dentistry, Swat. The study will recruit 344 patients aged above 10 and below 60 years, with permanent first molars indicated for RCT and meeting specific clinical and radiographic criteria. Participants will be randomly allocated into two groups: one receiving single-visit RCT and the other receiving multiple-visit RCT. Pain and flare-up incidence will be evaluated using the Visual Analog Scale (VAS) and swelling grading criteria at 6, 24, and 48 hours post-treatment. The primary outcome is the frequency of endodontic flare-ups requiring additional intervention. The study also examines the role of occlusal reduction in managing postoperative discomfort. Data will be analyzed using SPSS v23 with chi-square and Fisher's exact tests to compare outcomes. The findings aim to inform evidence-based protocols for endodontic treatment in the local population.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to compare the frequency of endodontic flare-ups following single-visit versus multiple-visit root canal treatment in patients presenting to Saidu College of Dentistry, Swat. An endodontic flare-up is defined as a significant postoperative complication characterized by unexpected severe pain and/or swelling occurring within hours to a few days after treatment and requiring unscheduled clinical intervention. The study will include 344 patients aged above 10 and below 60 years, with deep caries and symptomatic irreversible pulpitis or symptomatic apical periodontitis in permanent first molars. All selected teeth will have complete root formation and periapical radiolucencies not exceeding 3x3 mm. Patients with systemic diseases, pregnancy, current or recent use of antibiotics, NSAIDs or corticosteroids, facial cellulitis, severe mobility, frank pus discharge, or significant root resorption will be excluded. The sample size is calculated using WHO sample size calculator with 80% power, 5% margin of error, and expected flare-up proportions of 18.3% for single-visit and 8.1% for multiple-visit groups based on prior research. Patients meeting inclusion criteria will be selected through purposive non-probability sampling and randomly assigned into two groups (single-visit and multiple-visit) using a lottery method. All patients will undergo a standardized treatment protocol including local anesthesia with 2% lidocaine and 1:100,000 epinephrine, rubber dam isolation, access preparation, canal irrigation with 5.25% sodium hypochlorite, and biomechanical preparation using ProTaper Universal rotary files. Working length will be determined using a Woodpecker apex locator and confirmed with radiographs. Apical patency will be maintained using a #10 K-file, and the apical width will be prepared three sizes larger than the initial binding file.

In the single-visit group, cleaning, shaping, and obturation will be completed in the same appointment, followed by restoration with light-cured glass ionomer cement. In the multiple-visit group, cleaning and shaping will be completed in the first appointment with medicament placement, and obturation will be performed in a subsequent visit. All canals will be obturated using the cold lateral compaction technique with gutta-percha and Kerr Sealapex sealer. After treatment, a final periapical radiograph will be taken. Postoperative pain will be assessed using the Visual Analog Scale (VAS) at 6, 24, and 48 hours post-treatment. Swelling will be graded on a 0-3 scale. A flare-up will be recorded if the patient reports pain ≥7 on the VAS or swelling grade ≥2 requiring analgesics or emergency care. Patients will be contacted via phone for pain monitoring, and instructed to report any sudden worsening of symptoms. Data will be recorded in a structured proforma.

The primary outcome measure is the incidence of endodontic flare-ups within 48 hours post-treatment. Secondary outcomes include postoperative pain intensity and need for unscheduled care. Data analysis will be conducted using SPSS v23. Mean and standard deviation will be calculated for continuous variables like age, and frequency and percentages for categorical variables like gender and flare-up incidence. The chi-square test will be used to compare flare-up rates between groups. Stratification will be done by age and gender to identify effect modifiers, and post-stratification chi-square or Fisher's exact test will be used as appropriate. A p-value of <0.05 will be considered statistically significant. The study aims to address the current gap in local literature regarding endodontic flare-ups in the Khyber Pakhtunkhwa population and evaluate the effectiveness of treatment protocols for better pain management in routine dental practice.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group >10 years with deep caries approximating pulp on radiograph and indicated for a root canal treatment.
* Proper bone support.
* No evidence of severe mobility/discharge of frank pus
* Radiographically tooth indicated for root canal treatment.
* Permanent first molars with periapical radiolucency not exceeding 3 mm × 3 mm in size.
* Complete root formation.
* Teeth in which the initial master file (K-File)binds at the apex were of ISO size 45 or less.

Exclusion Criteria:

* Tooth/teeth with extensive periodontal pathology/ periapical radiolucency.
* Teeth with evidence of internal or external root resorption involving more than one third of the root length.
* Children with facial cellulitis or significant extraoral swelling.
* Patients with any systemic diseases.
* Patients who had been taking Antibiotics ,nonsteroidal anti-inflammatory drugs, corticosteroids at time of treatment.
* Pregnant patients

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of endodontic flare-ups | With in 48 hours after root canal treatment
  Flare-up defined as severe postoperative pain (VAS score ≥ 7) and/or swelling requiring unscheduled dental intervention, excluding pre-existing conditions

CONTACTS AND LOCATIONS:
Overall Officials: Warisha Ubaid, Principal Investigator — Saidu College of Dentistry Swat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This randomized controlled trail compares the incidence of endodontic flare ups (pain/swelling)between single visit and multiple visit root canal treatment.This study conducted at Saidu College of Dentistry,Swat, monitors patients over 6months . — http://prsinfo.clinicaltrials.gov/
- Available data/document: Study Protocol — http://www.scd.edu.pk